CLINICAL TRIAL: NCT00391586
Title: INST 0601C: A Non-Randomized Phase II Protocol of Erlotinib for Patients With Newly Diagnosed, Advanced Non-Small Cell Carcinoma of the Lung
Brief Title: Erlotinib and Standard Platinum-Based Chemotherapy for Newly Diagnosed, Advanced Non-Small Cell Carcinoma of the Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0601C; NCI-2012-01264 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: erlotinib; NSCLC; chemotherapy; platinum; lung; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Platinum Compounds; Paclitaxel; Platinum; Docetaxel; Vinorelbine; Pemetrexed; Irinotecan; Etoposide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib followed by chemotherapy (Experimental): Erlotinib: 150 mg orally once daily,
  Platinum-based chemotherapy regimen selections include:
  Carboplatin (Carbo) area under the curve (AUC) 6, or cisplatin (Cis) 60-100 mg/m2, day (D)1, administered with one of the following:
  1. Docetaxel 75 mg/m2, D1
  2. Docetaxel 35 mg/m2, D1,8,15
  3. Paclitaxel 200-225 mg/m2, D1
  4. Paclitaxel 80-100 mg/m2, D1,8,15
  Carbo AUC 5-6, or Cis 60-100 mg/m2, D1, administered with one of the following:
  1. Etoposide 100 mg/m2 D1-3
  2. Etoposide 200 mg/m2 orally D1-3
  3. Pemetrexed 500 mg/m2, D 1
  4. Irinotecan 50 mg/m2 D1,8,15
  Other regimens:
  1. Gemcitabine 1000 mg/m2-1250 mg/m2, D1,8 + Carbo AUC 6, or Cis 60-100 mg/m2, D1 or 8
  2. Vinorelbine 25 mg/m2 D1,8 + Carbo AUC 5, or Cis 80 mg/m2 D1
  Interventions: Drug: Erlotinib; Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered for at least 2 cycles (6 weeks) and for a maximum of 8 months.
  Upon progression or intolerance to erlotinib, standard of care platinum-based chemotherapy (per the choice of the treating physician) is administered every 3 weeks. Physicians can adjust dose, schedule, or supportive care to the benefit of the patient
  Other Names: Tarceva; OSI-774
Drug: Platinum-based chemotherapy — Intravenous chemotherapy combination per physician discretion every 3 weeks for at least 2 cycles
  Other Names: paclitaxel + platinum; docetaxel + platinum; vinorelbine + platinum; pemetrexed + platinum; irinotecan + platinum; etoposide + platinum; gemcitabine + platinum

SUMMARY:
This study was conducted to compare the activities of erlotinib to that of intravenous, platinum-based therapy in the treatment of non-small cell lung cancer (NSCLC). The goal of this trial was to demonstrate clinical equivalence of erlotinib to platinum-based frontline therapy, compared to historical controls.

DETAILED DESCRIPTION:
To compare the activities (the progression-free survival, the incidence and severity of toxicities, and reversibility of toxicities) of erlotinib to that of platinum-based therapy in NSCLC. A sequential therapy design has been chosen such that all patients will receive any potential benefits of both platinum-based and erlotinib therapy, without compromising survival by denying anyone potential therapy. With this design, progression-free survival will be tracked by treatment received. However, data will be generated which will show the safety and efficacy of erlotinib in the frontline setting (alone and with historical comparison to platinum-based therapy), as well as the potential safety and activity of platinum-based therapy in the "second-line" (post-erlotinib) setting. This should allow for the demonstration of the relative median time to progression, objective response and clinical benefit rates, overall survival, and safety and tolerability of erlotinib and platinum-based therapy in both the frontline and second-line settings in NSCLC. Also, in this fashion, the treatments serve as controls for each other, as well as being compared to historical controls; in the first line treatment portion, the platinum-based regimens serve as the historical control, while in the second-line setting, erlotinib serves as the historical control arm.

ELIGIBILITY:
Inclusion Criteria:

* Prior chemotherapy will be allowed for other invasive malignancies, provided at least five years has elapsed since the completion of therapy and enrollment on this protocol. No prior chemotherapy for metastatic non-small cell lung cancer (NSCLC) will be allowed. Prior adjuvant or neoadjuvant chemotherapy for NSCLC will be allowed, provided at least six months have elapsed from the last dose of chemotherapy to the documentation of relapsed disease.

Baseline laboratory values (bone marrow, renal, hepatic):

* Adequate bone marrow function:

  * Absolute neutrophil count >1000/µL
  * Platelet count >100'000/µL
* Renal function:

  * Serum creatinine < 2.0 mg %
* Hepatic function:

  * Bilirubin <1.5x normal
  * Serum calcium < 12 mg/dl

Other Eligibility Criteria:

* Signed Informed Consent
* Eastern Cooperative Oncology Group (ECOG)/Zubrod/Southwest Oncology Group (SWOG) Performance Status <2 (Karnofsky Performance Status > 70%)
* Life expectancy > 8 weeks
* Male or female' age >18 years
* Patients of childbearing potential must be using an effective means of contraception.
* Histologic diagnosis of NSCLC that is advanced and cannot be treated adequately by radiotherapy or surgery; or metastatic disease

Exclusion Criteria:

* Prior therapy with an epidermal growth factor receptor inhibitor, including erlotinib, gefitinib, and cetuximab, as well as any investigational HER-1 inhibiting agent
* Pregnant or lactating females
* Myocardial infarction or ischemia within the 6 months before Cycle 0' Day 0
* Uncontrolled' clinically significant dysrhythmia
* History of prior malignancy within the prior five years, with the exception of non-melanoma carcinomas of the skin, and carcinoma in situ of the cervix
* Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* Uncontrolled metastatic disease of the central nervous system (previously treated, stable disease is allowable on this protocol)
* Radiotherapy within the 2 weeks before Cycle 1' Day 1
* Surgery within the 2 weeks before Cycle 1' Day 1
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-07; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennie V Jones, MD, Principal Investigator — University of New Mexico
Locations (5):
- United States (5):
  - Lovelace Medical Group, Albuquerque, New Mexico
  - Hematology Oncology Associates NM, Albuquerque, New Mexico
  - Presbyterian Medical Group, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico

REFERENCES:
- See also: UNM CRTC Homepage — http://cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 07/13/2006 and ended 02/09/2009. All patients were recruited through medical clinics in New Mexico, USA.
Groups:
- Erlotinib Followed by Chemotherapy: Erlotinib at 150 mg orally per day for at least 2 cycles (6 weeks) and for a maximum of 8 months. Upon progression or drug intolerance, this is followed by standard of care platinum-based chemotherapy selected by the treating physician, every 3 weeks for at least 2 cycles
Period: Overall Study
Arm/Group | Erlotinib Followed by Chemotherapy
Started | 45
Received First-line Erlotinib | 43 (These patients received at least one dose of on-study first-line erlotinib)
Received Platinum-based Chemotherapy | 10 (Total number of patients who received platinum-based chemotherapy after erlotinib treatment)
Completed | 21 (These patients received at least 2 cycles of erlotinib)
Not Completed | 24
Not completed — Progressive disease | 13
Not completed — Adverse Event | 5
Not completed — Physician Decision | 2
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: These are patients who received at least one dose of on-study erlotinib
Arm/Group | Erlotinib Followed by Chemotherapy
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 68 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Time Frame: 5 years
Population: This study was terminated early; no results are available. The number of patients who completed treatment and therefore the number of evaluable patients was too low to accurately calculate endpoints.
Arm/Group | Erlotinib Followed by Chemotherapy
Number analyzed (Participants) | 0

2. Primary Outcome: Toxicity Profile
Description: Toxicities are assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 3.0. Toxicities are reported as the number of patients who experienced grade 3 or grade 4 adverse events after receiving at least one dose of on-study treatment.
Time Frame: 28 days after last on-study treatment
Measure: Number; unit: participants
Arm/Group | Erlotinib Followed by Chemotherapy
Number analyzed (Participants) | 43
participants
  Acne | 1
  Anorexia | 1
  Confusion | 1
  Dehydration | 1
  Diarrhea | 2
  Dyspnea | 3
  Fatigue | 8
  Nasal hemorrhage | 1
  Insomnia | 1
  Kidney pain | 1
  Lymphocyte count decreased | 1
  Muscle weakness | 1
  Neutrophil count decreased | 2
  Desquamating rash | 1
  Syncope | 1
  Thrombosis (clotting) | 1

ADVERSE EVENTS:
Time Frame: Patients are assessed for toxicity/adverse events for 28 days after completion of the last course of any on-study therapy.
Arm/Group | Erlotinib Followed by Chemotherapy
Serious Adverse Events (participants affected / at risk) | 5/43
Other Adverse Events (participants affected / at risk) | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib Followed by Chemotherapy (N=43)
Glucose intolerance (Endocrine disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Clotting) (Blood and lymphatic system disorders) | 1 (1)
Ear, nose, and throat examination abnormal (General disorders) | 1 (1) — Sore throat, dysphagia (trouble swallowing), and painful lymph node
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib Followed by Chemotherapy (N=43)
Fatigue (General disorders) | 13 (25)
Fever (General disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 9 (13)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 7 (9)
Anorexia (loss of appetite) (Gastrointestinal disorders) | 8 (13)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 9 (16)
Nausea (Gastrointestinal disorders) | 9 (9)
Taste alteration (Gastrointestinal disorders) | 7 (9)
Vomiting (Gastrointestinal disorders) | 4 (5)
Dizziness (Nervous system disorders) | 3 (3)
Insomnia (Nervous system disorders) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Chest pain (General disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pleural effusion (Fluid collection in lung lining) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No